CLINICAL TRIAL: NCT02387086
Title: A Phase III, Multi Center, Randomized, Placebo Controlled Study to Evaluate the Efficacy of the Combination Gefitinib With Thalidomide in Patients With Locally Advanced and Metastatic Non-Small-Cell-Lung-Cancer With EGFR Mutation
Brief Title: Gefitinib Combined With Thalidomide to Treat NSCLC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bai Jun (Other)
Responsible Party: Sponsor-Investigator, Bai Jun, Doctor, Shaanxi Provincial People's Hospital
Organization: Shaanxi Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GELI
Record Dates: First submitted 2015-03-03; First posted 2015-03-12 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: NSCLC
Keywords: gefitinib; thalidomide; NSCLC; EGFR mutation
MeSH Terms: interventions — Thalidomide; Gefitinib; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A:gefitinib and thalidomide/aspirin (Experimental): intervention: drug: gefitinib and thalidomide/aspirin: gefitinib will be administered at 250mg QD continuously; thalidomide will be administered at 100mg QD at night continuously; aspirin will be administered at 100mg QD continuously;
  Interventions: Drug: Thalidomide; Drug: Gefitinib; Drug: Aspirin
- B:Placebo (Placebo Comparator): intervention: drug: gefitinib and placebo/aspirin: gefitinib will be administered at 250mg QD continuously; placebo will be given to patients in the same way as the thalidomide; aspirin will be administered at 100mg QD continuously;
  Interventions: Drug: placebo; Drug: Gefitinib; Drug: Aspirin

INTERVENTIONS:
Drug: Thalidomide
  Arms: A:gefitinib and thalidomide/aspirin
Drug: placebo
  Arms: B:Placebo
Drug: Gefitinib
Drug: Aspirin

SUMMARY:
The purpose of this study is to determine whether thalidomide can improve the effectiveness of the gefitinib in NSCLC patients with EGFR mutations.

DETAILED DESCRIPTION:
Primary Objective:

To determine the 1 year progression-free survival(PFS) rate of the combination of thalidomide with gefitinib in patients who harbors EGFR mutations.

Secondary Objectives:

1. To evaluate the objective response rate and 2 years overall survival of this combination therapy;
2. To evaluate the safety and tolerability of this combination therapy;
3. To acquire preliminary data regarding the effects of thalidomide on interleukin-2 level in serum.

Treatment will be administered on an outpatient basis. Thalidomide starting at a dose of 50mg QD at night. After one week, increase the dose to 100mg QD at night.

Aspirin will be administered at 100mg QD continuously. Gefitinib will be administered at 250mg QD continuously. Maintenance Therapy patients responding to this therapy will be maintained with gefitinib、thalidomide and aspirin.

Duration of Therapy

In the absence of treatment delays due to adverse events, treatment may continue until one of the following criteria applies:

1. Disease progression,
2. Intercurrent illness that prevents further administration of treatment,
3. Unacceptable adverse events(s),
4. Patient decides to withdraw from the study, or
5. General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be NSCLC confirmed by Histological or cytological;
* The NSCLC harbors EGFR-mutation and are previously untreated
* Patient must have measurable lesion and in stage IIIB or IV disease (includes M1a, M1b stages or recurrent disease) (according to the 7th edition of the tumor node metastasis (TNM) classification system).
* Patients be age >18 years and < 75 years.
* Patients must have a Life Expectancy of greater than 12 weeks.
* Patients must have an ECOG performance status 0 to 2.
* Patients must have normal organ and marrow function as defined below, within one week prior to randomization: absolute neutrophil count>1,500/mL platelets>100,000/mL total bilirubin: within normal institutional limits AST/ALT<2.5X institutional upper limit of normal creatinine≤1.5X institutional upper limit of normal urine dipstick for proteinuria of < less than 1+. If urine dipstick is > 1+ then a 24 hour urine for protein must demonstrate <500mg of protein in 24 hours to allow participation in the study.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Patients must have an international normalized ratio (INR) < 1.5 and a partial thromboplastin time (PTT) no greater than upper limits of normal within 1 week prior to randomization.
* Patients with a history of hypertension must be well-controlled (<150 systolic/<100 diastolic) on a stable regimen of anti-hypertensive therapy.
* Patients must be able to swallow tablets.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
* Patients receiving therapeutic anticoagulation. Prophylactic anticoagulation of venous access devices is allowed provided Section 3.10 is met. Caution should be taken on treating patients with low dose heparin or low molecular weight heparin for DVT prophylaxis during treatment with bevacizumab as there may be an increased risk of bleeding.
* Patients cannot administer aspirin for the risk of bleeding or having stomach ulcers.
* Prior use of chemotherapy.
* Patients receiving immunotherapy, hormonal-therapy and or radiotherapy within 2 weeks prior to entering the study. Note: Those who have not recovered from adverse events due to these agents administered will be considered ineligible.
* Patients receiving any other investigational agents.
* Patients with uncontrolled brain metastasis. Note: Patients with brain metastases must have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks, and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to thalidomide、gefitinib and aspirin or other agents used in the study are excluded.
* Women that are pregnant or breastfeeding Note: Pregnant women are excluded from this study because the agents used in this study may be teratogenic to a fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with thalidomide, breastfeeding women are also excluded from this study.
* HIV-positive Patients that are on combination antiretroviral therapy due to the potential for lethal infections when treated with marrow-suppressive therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 1 year
  one year progression-free survival of the patients

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  the Objective Response Rate
Overall Survival (OS) | 2 years
  2 years Overall Survival

OTHER OUTCOMES:
IL-2 level | 2 years
  IL-2 level in serum of patients

CONTACTS AND LOCATIONS:
Overall Officials: Jun Bai, Principal Investigator — Shaanxi Provincial People's Hospital